CLINICAL TRIAL: NCT05539703
Title: The Effectiveness of Offering a 2nd Booster Dose of COVID-19 Vaccine on Preventing Severe COVID-19; A Register-based Randomized Trial (RRCT)
Brief Title: Trial of 2nd Booster Dose of COVID-19 Vaccine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not get the necessary approvals in time.
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REK 476603
Record Dates: First submitted 2022-09-13; First posted 2022-09-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The trial is designed as a register-based randomized trial. The investigators will draw a random sample from the whole population aged 45-64 years, which will constitute the intervention group and will receive a personal offer to receive a 2nd booster dose of a COVID-19 vaccine in their municipality. The rest of the population aged 45-64 will receive no such offer or information and will serve as control group. The random sample will be defined by drawing a set of birth dates. This allows the investigators to identify persons in the intervention group directly in the Norwegian Preparedness Register for COVID-19 without identifying them individually, since personal identification numbers are encrypted in this database. The random sample will receive the offer of vaccination either (i) via Helsenorge (National online health services in Norway) , or (ii) directly from their municipality.
Who Masked: Outcomes Assessor
Masking Description: We will, to the extent feasible, mask the data analysts to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention groups: Invitation to get 2nd booster (Experimental): Participants in the intervention group will receive an invitation to get a 2nd COVID-19 booster dose. Those who accept the invitation to be vaccinated will receive the vaccine through their municipality's vaccination service.
  Interventions: Other: Invitation to get a 2nd booster dose of COVID-19 vaccine
- Control group: No invitation to get 2nd booster (No Intervention): The control group will receive no intervention.

INTERVENTIONS:
Other: Invitation to get a 2nd booster dose of COVID-19 vaccine — Participants in the intervention group will receive an invitation to get a 2nd COVID-19 booster dose. Those who accept the invitation to be vaccinated will receive the vaccine through their municipality's vaccination service.
  Arms: Intervention groups: Invitation to get 2nd booster

SUMMARY:
Background Recent studies indicate that a 2nd booster dose is associated with lower risk of severe COVID-19. The studies are based on Israeli registry data, comparing outcomes among individuals who have taken the booster, or not. Interpreting the findings from such non-experimental studies is challenging - there are likely systematic differences between those who accept the offer to take a booster dose, and those who do not.

Aim Determine the effect of offering vaccination with a 2nd COVID-19 booster dose on severe COVID-19, measured by hospitalization and death caused by COVID-19.

Methods Intervention group: A random sample drawn from the whole population aged 45-64 years with 3 doses of COVID-19 vaccine will receive a personal offer to receive the 4th dose of a COVID-19 vaccine in their municipality.

Control group: The rest of the population aged 45-64 with 3 doses, who will receive no such offer.

Randomization: The investigators will draw a set of birth dates - can then see who is in the intervention group in Beredt C19 (Norwegian emergency preparedness register for COVID-19) without identifying them individually (personal identification numbers are encrypted).

Primary outcome: Hospitalization or death caused by COVID-19 in a period of 10 weeks after invitations are sent.

Sample size calculations: 300 000 individuals in the intervention group, assuming risk of the primary outcome is at least 15% lower in the intervention group. (The investigators expect a large proportion NOT to accept the invitation to take the vaccine).

DETAILED DESCRIPTION:
Background and rationale

Several studies suggest a waning of COVID-19 vaccines' effectiveness over time, raising the question of whether booster doses should be offered to maintain protection against severe COVID-19.

Studies of the effectiveness of taking one booster dose, which for most people corresponds to a third vaccine dose, have shown promising results. Similarly, three recent studies examining the effectiveness of a 2nd booster dose found that the 2nd booster was associated with lower risk of severe COVID-19. All these studies are based on data from Israeli registries, comparing outcomes among individuals who have taken the booster, or not. Interpreting the findings from such non-experimental studies is challenging since there are likely systematic differences between those who accept the offer to take a booster dose, and those who do not. So called "healthy vaccinee bias" implies that those who take the vaccine are healthier than those not taking the vaccine. The opposite, however, may also be true: Those who perceive themselves to be more at risk may be more prone to accept the offer of vaccination. A related type of bias is the "premature efficacy bias" which is observed in many observational studies within one to two weeks after vaccination, probably due to people refraining from taking the vaccine if they suspect that they have already been infected. Comorbidities or socio-economic factors that are not adequately controlled for can also lead to biased results. The conventional approach to minimizing the risk of bias in effectiveness studies is to conduct a randomized trial - if feasible.

The future of the COVID-19 pandemic is unknown. In Norway, a large winter wave driven by the omicron variant of SARS-CoV-2 is receding after more than half the population has been infected. The vaccination coverage in the Norwegian population is also very high.

In the autumn of 2022, a new wave of infections may start due to waning immunity, and/or the emergence of a new variant.

Either way, vaccination will be the most important tool to reduce the risk of severe disease in individuals. Based on previous experiences and the available data, it is likely that health authorities in Norway (and probably other European countries) will offer or even recommend a 2nd booster dose (the fourth dose) to those who are aged 65 years and above. For those who are younger and therefore at lower risk of severe COVID-19, the value of a 2nd booster is less clear, making it difficult to decide for or against offering a 2nd booster to this group.

The investigators therefore propose to conduct a register-based randomized trial (RRCT) to provide evidence for the effects of offering a 2nd booster (a fourth dose) in the age group 45-64 years.

Objectives Our primary objective is to determine the effect of offering vaccination with a COVID-19 booster dose on severe COVID-19, measured by hospitalization and death caused by COVID-19.

Our secondary objective is to determine the effects (intended and unintended) of offering vaccination with a COVID-19 booster dose on the use of health care services, prescription medication related to COVID-19, and on SARS-CoV-2 infection rate.

Trial design The trial is designed as a register-based randomized trial. The investigators will draw a random sample from the whole population aged 45-64 years, which will constitute the intervention group and will receive a personal offer to receive a 2nd booster dose of a COVID-19 vaccine in their municipality. The rest of the population aged 45-64 will receive no such offer or information and will serve as control group. The random sample will be defined by drawing a set of birth dates. This allows the investigators to identify persons in the intervention group directly in the Norwegian Preparedness Register for COVID-19 without identifying them individually, since personal identification numbers are encrypted in this database. The random sample will receive the offer of vaccination either (i) via Helsenorge (National online health services in Norway) through a survey tool available to the Norwegian Institute of Public Health, or (ii) directly from their municipality (to be determined).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 and 64 years
* Registered in the Norwegian national population register
* Have received three doses of a COVID-19 vaccine, with the last dose received at least four months ago.
* Have not previously been offered or recommended a 4th dose for medical reasons

Exclusion Criteria:

* Persons who have already been offered a 4th COVID-19 vaccine dose.
* Persons in whom COVID-19 vaccination is contraindicated as per the vaccines' Summary of Product Characteristics (SPC).

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Severe COVID-19 | To be decided, but no more the 3 months
  Hospitalization or death caused by COVID-19 starting on day 22 after the invitation is sent to the intervention group.

SECONDARY OUTCOMES:
Hospitalization or death | 10 weeks
  Hospitalization or death from all causes
Health care utilization | 10 weeks
  Health care utilization and use of prescription medication related to COVID-19
COVID-19 infection | 10 weeks
  Registered COVID-19 infection
Health care utilization related to potential side effects | 10 weeks
  Health care utilization related to potential side effects of the COVID-19 vaccine (e.g., myocarditis)
Infection, hospitalization or death | 12 months
  Infection, hospitalization or death in a period of 12 months starting from the date of receiving the 1st booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD MD, Study Director — Norwegian Institute of Public Health

IPD SHARING:
Plan to Share IPD: Yes
We intend to give full access to the full protocol and statistical code, to anyone who is interested. We also intend to share anonymised IPD to the extent possible within the existing legal framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We intend to make data available around six months after trial-start. The data will be available for at least 5-10 years.
Access Criteria: No criteria - anyone who is interested will be given access.